CLINICAL TRIAL: NCT03374826
Title: Non-invasive Axillary Lymph Node Staging in Breast Cancer With PET-MRI
Brief Title: PET-MRI for Axillary Staging in Node Negative Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL62441.068.17
Record Dates: First submitted 2017-11-28; First posted 2017-12-15 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Diseases
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dedicated axillary hybrid PET-MRI axilla (Experimental)
  Interventions: Diagnostic Test: Dedicated axillary hybrid PET-MRI

INTERVENTIONS:
Diagnostic Test: Dedicated axillary hybrid PET-MRI — All clinically node negative patients will undergo a hybrid PET-MRI axilla preoperatively, followed by breast surgery and SLNB.

SUMMARY:
Axillary lymph node status is an important prognostic factor for patients with breast cancer. After breast cancer diagnosis, current nodal staging consists of axillary ultrasound (US) combined with tissue sampling when deemed necessary. In case of positive axillary lymph nodes, patients will undergo axillary lymph node dissection (ALND). In case of no suspicious axillary lymph nodes (i.e. clinically node negative patients), patients will undergo sentinel lymph node biopsy (SLNB). This surgical nodal staging is accompanied by co-morbidity. In theory, if non-invasive imaging can evaluate the lymph node status accurately, a node negative patient would no longer have to undergo axillary surgery. Since MRI is suitable for soft tissue imaging and PET has the advantage of showing increased metabolic uptake in lymph node metastases, a combination of these techniques in hybrid PET/MRI would be highly desirable. If dedicated axillary hybrid PET/MRI is equally accurate to SLNB for the detection of negative axillary lymph nodes, work-up could be more efficient by bypassing SLNB. However, the accuracy of dedicated axillary hybrid PET/MRI needs to be compared with the pathological outcome of SLNB (gold standard) first.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient with histologically confirmed breast cancer and clinically confirmed negative lymph nodes in the axilla, scheduled to undergo SLNB
2. Patients who are willing and able to undergo the study procedures
3. The patient has provided personally written informed consent

Exclusion Criteria:

1. Patients treated with neoadjuvant systemic therapy prior to axillary nodal staging
2. Patients with clinically positive axillary lymph nodes
3. Age < 18 years
4. Inability to provide informed consent
5. Pregnancy
6. Weight >100 kg (because of the format of the PET/MRI scanner)
7. General contraindications for MRI (such as pacemaker, aneurysm clips, metallic device in their body, severe claustrophobia) or PET (i.e. known allergy to 18F-FDG)
8. Hyperglycaemia (> 11 mmol/L) at the time of 18F-FDG injection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of dedicated hybrid PET/MRI | Participants will be followed from the moment of first outpatient clinic visit until final breast surgery, an expected average of 4 weeks
  Accuracy (sensitivity, negative predictive value (NPV) and false negative rate (FNR)) of dedicated axillary hybrid PET/MRI to exclude axillary lymph node metastases will be calculated.

SECONDARY OUTCOMES:
Accuracy of T2w MRI, DWI and Hybrid PET/MRI | Participants will be followed from the moment of first outpatient clinic visit until final breast surgery, an expected average of 4 weeks
  Accuracy (sensitivity, negative predictive value (NPV) and false negative rate (FNR)) of three MRI sequences (T2w, DWI and hybrid PET/MRI) to exclude axillary lymph node metastases will be calculated separately as well.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No